CLINICAL TRIAL: NCT01130662
Title: Phase I Open-Label Study of Decitabine in Combination With Midostaurin (PKC412) for Elderly (Age ≥ 60) Newly Diagnosed or Relapsed/Refractory Adult Patients With Acute Myeloid Leukemia
Brief Title: Combination of Decitabine and Midostaurin in Patients Older Than 60 With Newly Diagnosed or Relapsed Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12010; CPCK412AUS06T (Other: Novartis)
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; AML; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine Midostaurin combination (Experimental)
  Interventions: Drug: combination therapy using decitabine and midostaurin

INTERVENTIONS:
Drug: combination therapy using decitabine and midostaurin — Cohort 1:
  Decitabine 20mg/m2 IV daily on days 1-5 to be repeated every 28 days. Midostaurin 25mg bid days 8-21 of each cycle.
  Cohort 2:
  Decitabine 20mg/m2 IV daily on days 1-5 to be repeated every 28 days. Midostaurin 50mg bid days 8-21 of each cycle.
  Cohort 3:
  Decitabine 20mg/m2 IV daily on days 1-5 to be repeated every 28 days. Midostaurin 50mg bid x 28 days of each cycle.
  Other Names: Dacogen; PKC412

SUMMARY:
The purpose of this study is to determine the tolerated dose of the combination of decitabine and midostaurin as induction (first cycle of chemotherapy) and consolidation (additional chemotherapy once a patient goes into remission) in people greater than 60 years with newly diagnosed AML or adult patients with relapsed/refractory disease.

DETAILED DESCRIPTION:
The development of a primarily outpatient treatment option for AML that is also capable of providing significant disease control is a priority for most clinicians. To address the need for less toxic, more effective treatments for older patients with AML, the purpose of this Phase 1 single institution study is to evaluate the safety and efficacy of midostaurin and decitabine administered in combination.

Decitabine is an epigenetic modifier of gene expression that has been shown to be well-tolerated in this population at the dose schedule proposed in this study, with reasonable efficacy. Although its precise mechanism of action is incompletely understood, it is postulated to work by reactivating the expression of key tumor suppressor genes silenced in tumor cells by reversing a pattern of hypermethylation of promotor elements.

Midostaurin is an oral agent that has been shown to inhibit FLT3 kinase in preclinical in vitro and in vivo studies, as well as clinically in patients with both ITD and TKD FLT3 mutations (FLT3mut). Both directly and indirectly, midostaurin also potently inhibits multiple other molecular targets thought to be important for the pathogenesis of AML. These targets include VEGFR-1, a VEGF receptor; c-kit; H- and K-ras; as well as the multidrug resistant gene, MDR.

The addition of midostaurin to a decitabine regimen of previously established efficacy and tolerability will allow us to evaluate the hypothesis that two drugs that are believed to work through distinct mechanisms of action may act together to improve the responses of patients treated with decitabine alone, without significant additional toxicity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age with newly diagnosed AML that is not eligible for standard induction or ≥ 18 years of age with relapsed/refractory AML
* Histologically documented AML (except t(15;17)according to the World Health Association (WHO) criteria
* Karnofsky performance status ≥ 70
* Must have the following lab values:
* AST and ALT < or equal to 2.5 x Upper Limit of Normal (ULN)
* Serum Bilirubin < or equal to 2.5 x ULN
* Serum Creatinine < or equal to 2.5 x ULN
* Must give written informed consent
* Left ventricular ejection fraction ≥ 50%

Exclusion Criteria:

* Prior allogeneic, syngeneic, or autologous bone marrow transplant or stem cell transplant less than 2 months previously
* Uncontrolled active infection
* Known impairment of GI function or GI disease that may significantly alter the absorption of midostaurin
* Female patients who are pregnant or breast-feeding or adults of reproductive potential not using an effective method of birth control. Barrier contraceptives must be used throughout the study in both sexes. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of midostaurin. Women considered not of childbearing potential include any of the following: no menses for at least 5 years or menses within 5 years but amenorrheic for at least 2 months and luteinizing hormone (LH) and follicular stimulating hormone (FSH) values within normal range (according to definition of postmenopausal for laboratory used) or bilateral oophorectomy or radiation castration and amenorrheic for at least 3 months.
* Other known disease (except carcinoma in-situ) concurrent severe and/or uncontrolled medical condition (eg uncontrolled diabetes, cardiovascular disease including congestive heart failure, myocardial infarction within 6 months and poorly controlled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study.
* Impaired cardiac function including any of the following:
* Screening ECG with a QTc > 450 msec
* Congenital long QT syndrome
* History or presence of sustained ventricular tachycardia
* Any history of ventricular fibrillation or torsades de pointes
* Bradycardia defined as HR less than 50 bpm
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Myocardial infarction or unstable angina < 6 months prior to starting study drug
* CHF NY Heart Association class III or IV
* Ejection fraction < 50% assessed by MUGA or ECHO scan within 14 days of Day 1
* Known confirmed diagnosis of HIV infection or active viral hepatitis
* Received any investigational agent within 30 days prior to Day 1
* Any surgical procedure, excluding central venous catheter placement, bone marrow biopsy or other minor procedures (eg skin biopsy) within 14 days of Day 1
* Unwilling or unable to comply with the protocol
* Known malignant disease of the central nervous system
* Any pulmonary infiltrate including those suspected to be of infectious origin. In particular, patients with resolution of clinical symptoms of pulmonary infection but with residual pulmonary infiltrates on chest x-ray are not eligible until pulmonary infiltrates have completely resolved
* Patients with prior midostaurin (PKC412) treatment are excluded
* Patients receiving any other investigational agents or have received other investigational agents within 30 days of enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to midostaurin and/or decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine a tolerated dose of the combination of decitabine and midostaurin as induction and consolidation in patients ≥ 60 years with newly diagnosed AML not eligible for standard induction or adult patients with relapsed/refractory disease. | 3 months per patient

SECONDARY OUTCOMES:
Explore potential association between clinical response and FLT-3 status in patients treated in each cohort; assess toxicity of combination in each dosing cohort | 3 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Casey Williams, PharmD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Westwood Campus, Kansas City, Kansas, United States